CLINICAL TRIAL: NCT01020643
Title: Comparison of Closed-loop Control System of Propofol Versus Manual Control Using Bispectral Index for Controlled Sedation - a Pilot Study
Brief Title: Closed-loop Sedation of Propofol for Patients Undergoing Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Hemmerling (Other)
Responsible Party: Sponsor-Investigator, Thomas Hemmerling, MSc, MD, DEAA,, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-168-GEN
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Conscious Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- controlled sedation using propofol (Experimental)
  Interventions: Drug: controlled administration of propofol

INTERVENTIONS:
Drug: controlled administration of propofol — comparison of propofol sedation

SUMMARY:
The purpose of this study is to compare the administration of a standard anesthetic drug (propofol) using an automatic, expert-based system versus a manually controlled system by the anesthesiologist. In addition, the performance of the decision support system will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hip or knee replacement under spinal anesthesia

Exclusion Criteria:

* contraindication to spinal anesthesia
* allergies to any study drug

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Controller performance | 1 year

SECONDARY OUTCOMES:
fluid management | end of surgery
  fluid management manual versus guided

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hemmerling, MD, Principal Investigator — MUHC - MGH
Locations (1):
- MUHC - Montreal General Hospital, Montreal, Quebec, Canada